CLINICAL TRIAL: NCT04150289
Title: A Disease Registry Encompassing the Care of Patients With Multiple Myeloma on Panobinostat (RECOMM)
Brief Title: A Disease Registry Encompassing the Care Of Patients With Multiple Myeloma on Panobinostat
Acronym: RECOMM
Status: Completed | Type: Observational
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 20192475
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Farydak; panobinostat
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Farydak — non-interventional study

SUMMARY:
This study aims to describe current treatment patterns in the real-world setting among patients with multiple myeloma who are initiating treatment with (or changing treatment to) panobinostat and explore the associations with baseline patient characteristics, healthcare resource utilization, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* At least 18 years of age
* Clinical diagnosis of multiple myeloma that meets published diagnostic criteria
* Initiating panobinostat within 60 days of enrollment
* ECOG performance status 0-1
* Availability of documentation from the patient's medical records regarding previous myeloma treatment, response, and duration of response
* Willing and able to complete the PRO questionnaire

Exclusion Criteria:

* Diagnosed with any B-cell malignancy other than myeloma
* Estimated life expectancy <6 months
* Currently enrolled in any interventional clinical trial at study entry (note: patients who enroll in an interventional clinical trial after enrollment may remain in the registry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be any adult who is clinically diagnosed with multiple myeloma who is actively taking panobinostat.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 24 months
  Looking for patient reproted response to treatment with panobinostat

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - American Health Network Indiana, Indianapolis, Indiana
  - Southern Nevada Cancer Research Foundation and Optum Cancer Care, Las Vegas, Nevada
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists, Huntersville, North Carolina
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: No